CLINICAL TRIAL: NCT01215357
Title: Ecopipam Treatment of Pathological Gambling
Brief Title: Clinical Study to Determine if Ecopipam Can Reduce Urges to Gamble
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: Psyadon Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PSY201; NCT01198951 (obsolete NCT alias)
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2013-02

CONDITIONS: Pathological Gambling
Keywords: Pathological Gambling; ecopipam; Dopamine
MeSH Terms: conditions — Gambling | interventions — ecopipam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ecopipam (Experimental): Ecopipam is a selective antagonist of one the classes of dopamine receptor.
  Interventions: Drug: Ecopipam
- Placebo (Placebo Comparator): Placebo given first week of the study.
  Interventions: Drug: Ecopipam

INTERVENTIONS:
Drug: Ecopipam — 50mg tablets
  Other Names: PSYRX101; SCH 39166

SUMMARY:
This study is designed to test the hypothesis that ecopipam is able to reduce urges to gamble in patients diagnosed with Pathological Gambling.

DETAILED DESCRIPTION:
The purpose of this study is to determine if ecopipam is able to stop urges to gamble in patients diagnosed with Pathological Gambling. Nerves communicate with each other by releasing chemicals called "neurotransmitters". One of these neurotransmitters in the brain is called "dopamine". After dopamine is released by the nerve it "talks" to other nerves by interacting with receptors that are unique to that neurotransmitter. Ecopipam is a drug that selectively blocks one family of dopamine receptors. Some scientists believe that the urge to gamble is related to having too much dopamine in the brain. By blocking the receptors that dopamine uses, ecopipam may be able to relieve the urge to gamble.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be diagnosed with Pathological Gambling according to DSMIV criteria
* Subject must have at least 2 episodes of gambling behavior within the previous 2 weeks before screening
* Subject must have gambling urges of at least moderate intensity

Exclusion Criteria:

* Subjects must not have unstable medical illness or clinically significant abnormalities on lab tests, ECG, or physical exam
* Subjects with major depressive episode within the last 2 years
* Subjects with a history of attempted suicide
* Subjects with first degree relative with major depressive episode that resulted in hospitalization, attempted or completed suicide
* Subjects with a history of epilepsy or seizures
* Subjects with a myocardial infarction (heart attack) with in the last 6 months
* Subjects with a lifetime history of bipolar disorder, dementia, schizophrenia, or any psychotic disorder
* Subjects with current of recent DSM-IV diagnosis of substance abuse or dependence (with the exception of nicotine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Grant, MD, Principal Investigator — Univ. of Minnesota; Donald Black, MD, Principal Investigator — Iowa University; Timothy Fong, MD, Principal Investigator — University of California, Los Angeles; Marc Potenza, MD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Carver College of Medicine, University of Iowa, Iowa City, Iowa
  - University of Minnesota School of Medicine, Minneapolis, Minnesota

REFERENCES:
- [Derived] Grant JE, Odlaug BL, Black DW, Fong T, Davtian M, Chipkin R, Kim SW. A single-blind study of 'as-needed' ecopipam for gambling disorder. Ann Clin Psychiatry. 2014 Aug;26(3):179-86. PMID 25166480
- See also: Psyadon Pharmaceutical's Website — http://www.psyadonrx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started Sept 2010 and finished June 2011
Pre-assignment Details: See exclusion criteria
Groups:
- Ecopipam (50 or 100 mg, as Needed): Patients were instructed to take a 50 mg tablet each time they had an urge to gamble. If that was ineffective, they were instructed to take a second 50 mg tablet. If that was ineffective, they were not allowed to increase the dose further.
Period: Overall Study
Arm/Group | Ecopipam (50 or 100 mg, as Needed)
Started | 34
Completed | 22
Not Completed | 12
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 9

BASELINE CHARACTERISTICS:
Groups:
- Ecopipam 50 or 100 mg, as Needed: Patients were instructed to take a 50 mg tablet of ecopipam when they had an urge to gamble. If no effect, then they could take a second 50 mg tablet. If still no effect, they were not permitted to take any more ecopipam.
Arm/Group | Ecopipam 50 or 100 mg, as Needed
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Statistically Significant (p<0.05) Decrease From Baseline in Yale Brown Obsessive Compulsive Scale Modified for Pathological Gambling
Description: This scale assesses the severity of gambling urges and gambling behaviors. The study anticipates that there will be a reduction in either or both of these assessments. The range is from a minimum of 0 to a maximum of 40, where zero means no gambling urges occurred.
Time Frame: Baseline and 6 weeks
Population: Patients completing all visits
Measure: Mean (Standard Deviation); unit: YBOCS score
Groups:
- Ecopipam 50 mg or 100 mg as Needed: Patients were instructed to take one 50 mg tablet of ecopipam when they had an urge to gamble. If this was effective, they should not take any more drug. If it was not effective, they were permitted to take a second 50 mg tablet of ecopipam. If this was effective, they should not take any more drug. If this was not effective, they were not permitted to take any additional ecopipam.
Arm/Group | Ecopipam 50 mg or 100 mg as Needed
Number analyzed (Participants) | 28
YBOCS score | 13.9 (8.79)

2. Secondary Outcome: Type, Frequency and Severity of Side Effects
Description: All side effects of the drug will be monitored and recorded
Time Frame: 6 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Statistically Significant Changes in the Gambling Symptom Assessment Scale
Description: It is expected that there will be decreases in this scale
Time Frame: 6 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Effects on the Clinical Global Impression
Description: Clinician's Global Impression is used assess severity and changes in clinical symptoms during and at the end of the study
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Ecopipam 50 or 100 mg, as Needed
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 13/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecopipam 50 or 100 mg, as Needed (N=34)
Sedation (Nervous system disorders) | 4 (4)
Anxiety (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Rhinorrhea (Eye disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This was an open label trial of ecopipam for the treatment of pathological gambling. A significant effect of drug treatment was demonstrated. These data need to be verified with a double-blind, placebo controlled trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less